CLINICAL TRIAL: NCT03469687
Title: 5 Year Clinical and Radiographic Follow-up of the Uncemented Symax Hip Stem in an International Study
Brief Title: Symax International Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Vejle Hospital (Other); Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 04-112
Record Dates: First submitted 2018-01-15; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-01

CONDITIONS: Hip Osteoarthritis; Prosthesis Durability
MeSH Terms: conditions — Osteoarthritis, Hip; Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symax uncemented hip stem (Other): The Symax hip stem is an uncemented design forged from Ti6Al4V alloy (Stryker EMEA). Primary mechanical stability is provided by anatomical metaphyseal geometry. The hip stem features a size dependent anteversion, neck length and offset, with a CCD angle of 128°. Secondary biological stability is accomplished by fast osseous integration due to the BONIT-HA coating on the metaphyseal part of the stem.
  Interventions: Device: Symax uncemented hip stem

INTERVENTIONS:
Device: Symax uncemented hip stem

SUMMARY:
The uncemented Symax hip stem is developed through optimization of the uncemented Omnifit hip stem. The Symax stem design combines an anatomical anteverted proximal geometry with a straight distal section. The proximal part is coated with a biomimetic hydroxyapatite (HA) coating for improved osseointegration to enhance load transfer and to minimize proximal bone loss. The distal part is treated with an anodization surface treatment in order to prevent distal bone apposition, which is expected to prevent distal loading and reduce proximal stress shielding. Aim of this study is to report mid-term clinical performance and evaluate whether the radiographic features are in line with the design principles of the Symax hip in an international clinical study with 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring uncemented primary total hip arthroplasty (osteoarthritis, avascular necrosis and/or post-traumatic arthritis), age between 18-70 years, BMI less or equal to 35.

Exclusion Criteria:

* Patients with bilateral hip complaints, impaired cognitive function and use of medication or illness influencing bone metabolism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-11-02 (Actual); Primary Completion 2010-10-11 (Actual); Study Completion 2010-10-11 (Actual)

PRIMARY OUTCOMES:
Change of Harris Hip Score (HHS) during follow-up | Preoperative HHS and postoperatively change in HHS at 6 months, 1 year, 2 years, 3 years and 5 years
  A hip specific functional score

SECONDARY OUTCOMES:
Radiographic evaluations | Immediately postoperative radiograhpic evaluation as baseline and changes in radiography at follow-up 6 months, 1 year, 2 years, 3 years and 5 years we evaluated the radiograhip evaluations again
  Radiographic evaluations per Gruen zone and comparison between two assessment teams

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] ten Broeke RH, Hendrickx RP, Leffers P, Jutten LM, Geesink RG. Randomised trial comparing bone remodelling around two uncemented stems using modified Gruen zones. Hip Int. 2012 Jan-Feb;22(1):41-9. doi: 10.5301/HIP.2012.9103. PMID 22383318
- [Result] ten Broeke RH, Alves A, Baumann A, Arts JJ, Geesink RG. Bone reaction to a biomimetic third-generation hydroxyapatite coating and new surface treatment for the Symax hip stem. J Bone Joint Surg Br. 2011 Jun;93(6):760-8. doi: 10.1302/0301-620X.93B6.24986. PMID 21586774
- [Derived] Kruijntjens DSMG, Kjaersgaard-Andersen P, Revald P, Leonhardt JS, Arts JJC, Ten Broeke RHM. 5-year clinical and radiographic follow-up of the uncemented Symax hip stem in an international study. J Orthop Surg Res. 2018 Jul 31;13(1):191. doi: 10.1186/s13018-018-0888-9. PMID 30064453